CLINICAL TRIAL: NCT01212263
Title: Clomiphene Citrate Co-treatment With Low Dose HP Urinary FSH vs. HP Urinary FSH Step-up Protocol for Clomiphene-citrate Resistant PCOS Anovulatory Infertility: Randomized Controlled Trial
Brief Title: Clomiphene Citrate (CC) Co-treatment With HP Urinary FSH vs HP Urinary FSH in CC-resistant PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura Integrated Fertility Center (Other)
Responsible Party: Principal Investigator, Mohamad Elsaid Ghanem, Dr, Mansoura Integrated Fertility Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MansouraIFC1
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Clomiphene resistance; ovulation induction; low dose uFSH; uFSH step-up protocol
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clomiphene Citrate plus HP uFSH (Experimental): Starting from the 2nd day of the cycle Clomiphene Citrate( CC)50 mg tablets are given in 100 mg daily dose for 5 days together with an low dose HP uFSH (half ampoule: 37.5 IU) given im daily for 8-10 days.
  Interventions: Drug: Clomiphine citrate plus low dose uFSH
- Step-up HP uFSH (Active Comparator): HP uFSH started in doses of half ampole (37.5 )IU daily from the 2nd day of cycle for 7 days ,then dose is stepped-up to one ampoule ( 75 IU) for 7 days then the one and a half amps (112.5) IU /day until follicular diameter reaches 18 mm mean diameter
  Interventions: Drug: Step-up HP u FSH

INTERVENTIONS:
Drug: Step-up HP u FSH — HP u FSH (Fostimone 75 IU ,IBSA Institut Biochimique SA-CH 6903 Lugano) in doses of 37.5 IU (half ampole) im /day statrted from second day of the cycle for 7 days ,then increased to 75 IU for another 7 days ,then to 112.5 IU (one and half ampoule) untilleading follicle mean diameter reaches 18 mm
  Arms: Step-up HP uFSH
Drug: Clomiphine citrate plus low dose uFSH — Clomiphene citrate 50 mg tab oral tablets(Clomid 50 mg tablets Global Napi , Egypt) two tablets(100 mg) /day are started from the 2nd day of cycle for 5 days togeteher with 37.5 IU HP uFSH (Fostimone 75 IU IBSA)/day for 8 days and may be extended to 10-12 days until leading follicle diameter reaches 18 mm
  Arms: Clomiphene Citrate plus HP uFSH

SUMMARY:
To test whether adding small doses of HP urinary FSH to standard regimen of clomiphene citrate in clomiphene resistant PCOS well yield better results in terms of better ovulation rate,lower follicle number, less consumption of HP urinary FSH,lower treatment cost , better pregnancy rate, lower multiple pregnancy rates compared with the exclusive use of HP urinary FSH in these cases.

DETAILED DESCRIPTION:
To test whether CC co- treatment with chronic low dose HP uFSH vs chronic low dose HP uFSH in CC resistant PCOS will yield better results in terms of ,ovulation rate, lower follicle number,lower HP uFSH dose ,better outcome in terms of pregnancy rates, better cost-effectiveness ratio, lower multiple pregnancy rates,lower cycle cancellation.

ELIGIBILITY:
Inclusion Criteria:

* CC resistant PCOS
* Infertile
* Females
* Age 18-38

Exclusion Criteria:

* Hyperprolactinaemia
* Cushing syndrome
* Adult onset adrenal hyperplasia
* Age >38
* Other infertility factors in the couple than PCOS: male factor,tubal factor,edometriosis

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
ovulation rate | 6 months
  IF CC Co-treatment with low dose step-up HP urinary(u)FSH results in similar or higher ovulation rate compared with step-up low dose HP uFSH

SECONDARY OUTCOMES:
Live birth rate | 6 months
  % of of cases that result in live birth > 20 weeks pregnancy
number of follicles sized 16 mm or more mean diameter in both ovaries at the time of hCG | 3 months
  To test if CC-co treatment with low dose HP uFSH results in lower number of follicles 16 mm mean diameter or more at time of triggerring ovulation compared with low dose HP uFSH
Endometrial thickness | 3 months
  Measuring endometrial thickness in mm in both study arms at the time of ovulation trigerring to see if there is difference
serum Estradiol(E2) | 3 months
  serum level of E2 is measured in both groups at the time of ovulation triggerring to test for differences
incidence of multiple pregnancy | 3 months
  To test if CC-co treatment with low dose HP uFSH results in lower or higher incidence of multiple pregnancies compared with low dose HP uFSH
costs per cycle | 3 months
  costs of drugs used to induce ovulation in each arm of the study in Egyptian pounds The cost of HP uFSH per cycle was calculated by multiplying the cost of a single IU with the mean number of FSH IU used per cycle. Add to this the cost of clomiphene citrate in the relevant arm
cost effectiveness ratio | 6 months
  The cost-effectiveness ratio is calculated multiplying the cost per cycle by the total number of cycles performed in each arm then dividing the result for the number of clinical pregnancies obtained in the arm during the trial.
clinical and biochemical predictors of response to treatment | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad E Ghanem, MD, Study Chair — Mansoura Integrated Fertility Center; Mohammad A Emam, MD, Study Director — Mansoura Integrated Fertility Center; Mohamad E Ghanem, MD, Principal Investigator — Mansoura Integrated Fertility Center
Locations (1):
- Mansoura Integrated fertility Center, Al Mansurah, Dekahlia, Egypt

REFERENCES:
- [Background] Palomba S, Falbo A, Zullo F. Management strategies for ovulation induction in women with polycystic ovary syndrome and known clomifene citrate resistance. Curr Opin Obstet Gynecol. 2009 Dec;21(6):465-73. doi: 10.1097/GCO.0b013e328332d188. PMID 19809318
- [Background] Gorry A, White DM, Franks S. Infertility in polycystic ovary syndrome: focus on low-dose gonadotropin treatment. Endocrine. 2006 Aug;30(1):27-33. doi: 10.1385/ENDO:30:1:27. PMID 17185789
- [Derived] Ghanem ME, Elboghdady LA, Hassan M, Helal AS, Gibreel A, Houssen M, Shaker ME, Bahlol I, Mesbah Y. Clomiphene citrate co-treatment with low dose urinary FSH versus urinary FSH for clomiphene resistant PCOS: randomized controlled trial. J Assist Reprod Genet. 2013 Nov;30(11):1477-85. doi: 10.1007/s10815-013-0090-2. Epub 2013 Sep 7. PMID 24014214